CLINICAL TRIAL: NCT04163185
Title: A Randomized, Double-blind, Single-dose, Placebo-controlled Study to Assess the Efficacy and Safety of AXS-07 (Meloxicam and Rizatriptan) for the Acute Treatment of Migraine in Adults
Brief Title: Initiating Early Control of Migraine Pain and Associated Symptoms
Acronym: INTERCEPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-07-303
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; AXS-07; Meloxicam; Rizatriptan
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXS-07 (Experimental): Taken once upon migraine
  Interventions: Drug: AXS-07 (MoSEIC meloxicam and rizatriptan)
- Placebo (Placebo Comparator): Taken once upon migraine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-07 (MoSEIC meloxicam and rizatriptan) — AXS-07 tablet taken once upon the earliest onset of migraine pain.
  Arms: AXS-07
Drug: Placebo — Placebo tablet taken once upon the earliest onset of migraine pain.
  Arms: Placebo

SUMMARY:
AXS-07 is an oral, investigational medicine consisting of MoSEIC meloxicam and rizatriptan, which is being developed for the acute treatment of migraine with or without aura in adults. AXS-07 tablets are formulated to provide an enhanced rate of absorption of meloxicam. This study is designed to evaluate the efficacy and safety of AXS-07 compared to placebo.

This is a randomized, double-blind, single-dose, placebo-controlled trial. Subjects who successfully complete the screening period and continue to meet all entry criteria will be randomly assigned to take one dose of either AXS-07 or placebo upon the earliest onset of migraine pain.

ELIGIBILITY:
Key Inclusion Criteria:

• Has an established diagnosis of migraine with or without aura.

Key Exclusion Criteria:

* Has previously received any investigational drug or device or investigational therapy within 30 days before Screening.
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Mobile, Alabama
  - Clinical Research Site, Colton, California
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Los Alamitos, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Santa Monica, California
  - Clinical Research Site, Spring Valley, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Hallandale, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lake City, Florida
  - Clinical Research Site, Lake Worth, Florida
  - Clinical Research Site, Ocoee, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, South Miami, Florida
  - Clinical Research Site, Sunrise, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Evanston, Illinois
  - Clinical Research Site, Louisville, Kentucky
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Waltham, Massachusetts
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Springfield, Missouri
  - Clinical Research Site, Albuquerque, New Mexico
  - Clinical Research Site, Manlius, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, High Point, North Carolina
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Mt. Pleasant, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Nashville, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Salt Lake City, Utah
  - Clinical Research Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Website — http://axsome.com

RESULTS

PARTICIPANT FLOW:
Groups:
- AXS-07: Taken once upon the onset of migraine
  AXS-07 (MoSEIC meloxicam and rizatriptan): AXS-07 tablet taken once upon the earliest onset of migraine pain.
- Placebo: Taken once upon the onset of migraine
  Placebo: Placebo tablet taken once upon the earliest onset of migraine pain.
Period: Overall Study
Arm/Group | AXS-07 | Placebo
Started (The Randomized Population included all subjects randomized to study drug.) | 152 | 150
Safety Population (The Safety Population included all subjects who received study drug.) | 140 | 143
ITT Population (The ITT Population consisted of all randomized subjects who had a qualifying migraine.) | 132 | 135
Completed | 140 | 143
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-07 | Placebo | Total
Number analyzed (Participants) | 140 | 143 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.58) | 41.4 (10.67) | 41.6 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 122 | 241
  Male | 21 | 21 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 7 | 8
  Black or African American | 18 | 17 | 35
  White | 118 | 116 | 234
  Multiple | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Headache Pain Freedom at Hour 2
Description: Absence of headache pain at Hour 2
Time Frame: Hour 2
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-07 | Placebo
Number analyzed (Participants) | 132 | 135
Participants | 43 | 22
Statistical Analysis 1: Comparison: AXS-07 vs Placebo; Test type: Superiority; p = 0.002, Chi-squared

2. Primary Outcome: Percentage of Subjects With Absence of Most Bothersome Symptom at Hour 2
Description: Absence of Most Bothersome Symptom, defined at the onset of migraine at Hour 2
Time Frame: Hour 2
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-07 | Placebo
Number analyzed (Participants) | 132 | 135
Participants | 58 | 36
Statistical Analysis 1: Comparison: AXS-07 vs Placebo; Test type: Superiority; p = 0.003, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected on or after the dosing date and included any new event or ongoing event that worsened in severity after the date of dosing. Adverse events were collected up to 5 days after the last study visit, up to 12 days per participant.
Description: Safety Population
Arm/Group | AXS-07 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/143
Other Adverse Events (participants affected / at risk) | 13/140 | 5/143
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AXS-07 (N=140) | Placebo (N=143)
Somnolence (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT04163185/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT04163185/SAP_002.pdf